CLINICAL TRIAL: NCT02171143
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP2409 Following a Single Intravenous Dose in Patients With Rheumatoid Arthritis on Methotrexate
Brief Title: A Dose Escalation Study to Assess Safety, Tolerability and Pharmacokinetics of ASP2409 Following a Single Intravenous Dose in Patients With Rheumatoid Arthritis on Methotrexate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2409-CL-0104
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Rheumatoid Arthritis; Pharmacokinetics of ASP2409
Keywords: ASP2409; Rheumatoid Arthritis; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ASP2409

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP2409 Dose Escalation (Experimental)
  Interventions: Drug: ASP2409
- Placebo Dose Escalation (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP2409 — intravenous (IV)
  Arms: ASP2409 Dose Escalation
Drug: Placebo — intravenous (IV)
  Arms: Placebo Dose Escalation

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of single, ascending, intravenous (IV) doses of ASP2409 in patients with Rheumatoid Arthritis (RA) on methotrexate (MTX) and to evaluate the pharmacodynamics (PD) of ASP2409.

DETAILED DESCRIPTION:
This is a dose-escalation study. Sequential cohorts of subjects will receive increasing doses of ASP2409 or matching placebo.

Subjects in all cohorts will stay confined in the unit for 3 days. All subjects will have scheduled outpatient visits and be followed for a minimum of 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject weighs at least 50 kg.
* Subject has a body mass index (BMI) of ≤ 35 kg/m2.
* Subject's 12-lead electrocardiogram (ECG) results are normal at Screening and Day -1 or, if abnormal, the abnormality is not clinically significant
* Female subject must be either:

  * Of non-childbearing potential:

    1. post-menopausal (defined as at least 1 year without any menses) prior to Screening, or
    2. documented surgically sterile or status post hysterectomy (at least 1 month prior to Screening).
  * Or, if of childbearing potential:

    1. must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1.
    2. must use two forms of birth control (at least one of which must be a barrier method) starting at Screening and throughout the Treatment and Observation Period, and for ≥ 120 days after final study drug administration.
    3. Acceptable forms include:

       1. Established use or oral, injected or implanted hormonal methods of contraception.
       2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
       3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) with spermicidal foam/gel/film/ cream/suppository.
* Female subject must not be breastfeeding at Screening or during the Treatment and Observation period and for ≥ 120 days after final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the Treatment and Observation period and for ≥ 120 days after final study drug administration.
* Male subject must not donate sperm starting at Screening and throughout the Treatment and Observation period and for at least ≥ 120 days after final study drug administration.
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continue throughout the Treatment and Observation period and for ≥ 120 days after final study drug administration.
* Subject has Rheumatoid Arthritis (RA) that was diagnosed according to the 1987 revised criteria of the American College of Rheumatology (ACR) ≥ 6 months prior to Screening.
* Subject meets the ACR 1991 revised criteria for Global Functional Status in RA, Class I, II or III at Screening.
* Subject MUST be on concomitant methotrexate (MTX):

  * for ≥ 3 months prior to study drug infusion, AND
  * at a stable dose (10 - 25 mg/week) for ≥ 28 days prior to study drug infusion and throughout the study.
* Subjects on the following medications must remain on a stable regimen: non-steroidal anti-inflammatory drugs (NSAIDs), selective cyclooxygenase-2 (COX-2) inhibitors, hydroxychloroquine (Plaquenil®), sulfasalazine, oral corticosteroids (≤ 10 mg of prednisone, or equivalent, daily) or low dose opioids (≤ 30 mg of oral morphine, or equivalent, daily) for

  ≥ 28 days prior to Screening and remain so throughout the Treatment and Observation Period. (The start of Plaquenil and sulfasalazine must be ≥ 2 months prior to study drug infusion.)
* Subject is highly likely to comply with the protocol and complete the study.

Exclusion Criteria:

* Subject has an ongoing clinically significant systemic disease such as uncompensated heart failure, uncontrolled diabetes mellitus, severe hepatic failure or severe pulmonary disease.
* Subject has a history of any malignancy except for adequately-treated, non-melanoma skin cancer and adequately-treated in-situ cervical cancer.
* Subject has a history of severe allergic or anaphylactic reactions.
* Subject has a history of consuming more than 14 units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/substance abuse within past 6 months prior to Screening (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits).
* Subject has a positive test for alcohol or drugs of abuse (excluding drugs prescribed to subject) at Screening or Day -1.
* Subject has/had a viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to Day -1.
* Subject has a past history of serious opportunistic infection.
* Subject is known positive for human immunodeficiency virus (HIV) antibody.
* Subject has a positive tuberculosis (TB) skin test or Quantiferon Gold test at Screening.
* Subject has a positive test for hepatitis C antibody, or positive test for hepatitis B surface antigen (HBsAg), or positive hepatitis B core antibody at Screening.
* Subject's laboratory test results at Screening:

  * alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST), are ˃ 2 times the upper limit of normal, AND/OR
  * are outside the normal limits and considered by the Investigator to be clinically significant with regard to the remaining per-protocol laboratory tests.
* Subject received any live or live attenuated vaccine within 30 days prior to study drug infusion.
* Subject received any systemic immunosuppressant agent, other than (MTX) or stable steroid regimen, within 2 months prior to study drug infusion.
* Subject has previously received any antibody or therapeutic biologic product within 56 days or 5 half-lives, whichever is longer, prior to study drug infusion.
* Subject has previously participated in any interventional clinical study or has received an experimental agent within 56 days or 5 half-lives, whichever is longer, prior to study drug infusion.
* Subject is participating in another clinical trial or has participated in another dose group of the current trial.
* Subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on Day -1.
* Subject has taken Orencia® (abatacept), Nulojix® (belatacept) or any other CTLA4-Ig molecule.
* Subject has any other condition which precludes the subject's participation in the trial.
* Subject has a history of prolonged QT syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ASP2409 concentration: Area under the concentration - time curve from time 0 up to the last quantifiable concentration (AUClast) | Days 1-8, Days 15, 22, 29, 43, 60, 90, and 120
Pharmacokinetics of ASP2409 concentration: Area under the concentration - time curve from time 0 extrapolated to infinity (AUCinf) | Days 1-8, Days 15, 22, 29, 43, 60, 90, and 120
Pharmacokinetics of ASP2409 concentration: Maximum concentration (Cmax) | Days 1-8, Days 15, 22, 29, 43, 60, 90, and 120
Safety assessed by adverse events | Up to 1 year
Safety assessed by laboratory tests | Up to 1 year
Safety assessed by electrocardiograms (ECGs) | Up to 1 year
Safety assessed by physical examinations | Up to 1 year
Safety assessed by vital signs | Up to 1 year
Safety assessed by anti-ASP2409 antibody formation | Up to 1 year

SECONDARY OUTCOMES:
Composite of pharmacokinetics of ASP2409 concentration: tmax, t1/2, Vz, Vss, CLtot | Days 1-8, Days 15, 22, 29, 43, 60, 90, and 120
  Time to attain Cmax (tmax), apparent terminal elimination half-life (t1/2), terminal phase volume (Vz), volume of distribution at steady-state (Vss), and total body clearance (CLtot)
Pharmacodynamics of ASP2409: CD86 receptor occupancy | Days 1-3, Days 5, 8, 15, 22, 29, 43, 60, and 90
  Cluster of Differentiation 86 (CD86), a co-stimulatory ligand on lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (10):
- United States (10):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - West Coast Clinical Trials, LLC, Costa Mesa, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Carolina Phase 1 Research, Raleigh, North Carolina
  - Community Research, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, LLC, Dallas, Texas
  - Texas Arthritis Research Center, San Antonio, Texas

REFERENCES:
- [Derived] Zhang W, Kernstock RM, Karrer EE, Cohen SB, Chindalore VL, Kivitz AJ, Blahunka PC, Delgado-Herrera L, Zeiher BG, Samberg NL, Garg JP. A Phase 1 Dose-Escalation Study of ASP2409, a Selective T-Cell Costimulation Inhibitor, in Stable Rheumatoid Arthritis Patients on Methotrexate Therapy. Clin Pharmacol Drug Dev. 2016 Jul;5(4):259-68. doi: 10.1002/cpdd.237. Epub 2016 Jan 8. PMID 27310327